CLINICAL TRIAL: NCT06683053
Title: Evaluation of the Use of Empagliflozin in Patients with Heart Failure with Preserved Ejection Fraction in a Cardiology Outpatient Department
Brief Title: Evaluation of the Use of Empagliflozin in Patients with HF with PEF in a Cardiology Outpatient Department
Acronym: ADDEMFEP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Conrado Roberto Hoffmann Filho (Network)
Responsible Party: Sponsor-Investigator, Conrado Roberto Hoffmann Filho, MD, Multidisciplinary Center for Specialized Education and Research Ltd.
Organization: Multidisciplinary Center for Specialized Education and Research Ltd. (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMEP
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Congestive Heart Failure (CHF)
Keywords: congestive heart failure; preserved ejection fraction; empagliflozin
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, randomized study comparing the efficacy and safety of empagliflozin at doses of 10 and 25 mg in patients with HFpEF. The Kansas City Cardiomyopathy Questionnaire (KCCQ TSS) will be applied at inclusion and 8 weeks post-intervention in the two groups. And the use of echocardiogram performed upon entering the study, with assessment of ventricular and atrial strain modalities, and being repeated at the end of the treatment period to try to detect possible differences between pre and post treatment with the proposed ISGLT2.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin 10 mg (Experimental): In this group the patients will receive the medication empagliflozin 10 mg
  Interventions: Drug: empagliflozin
- Empagliflozin 25 mg (Experimental): In this group the patients will receive the medication empagliflozin 25 mg.
  Interventions: Drug: empagliflozin

INTERVENTIONS:
Drug: empagliflozin — Comparing the benefits of both doses of empagliflozin (10 mg versus 25 mg) in terms of heart ejection fraction and quality of life.

SUMMARY:
This study aims to evaluate whether the use of a 25 mg dose of empagliflozin compared to the 10 mg dose used would bring additional benefits in the improvement outcomes of the Kansas City Cardiomyopathy Questionnaire (KCCQ SST), in the 6-minute walk test (6MWT) without causing significant side effects.

DETAILED DESCRIPTION:
This study aims to evaluate whether the use of a 25 mg dose of empagliflozin compared to the 10 mg dose used would bring additional benefits in the improvement outcomes of the Kansas City Cardiomyopathy Questionnaire (KCCQ SST), in the 6-minute walk test (6MWT) without causing significant side effects. Patients will be randomized and will receive one of the two doses of empagliflozin. All patients in both groups will be equally evaluated by the tests, before receiving the medication, and also 8 weeks after.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old.
* Echocardiogram with ejection fraction > 50%
* Patients must present at least one of the following items to be included in the study: Patients with a previous diagnosis of Heart Failure with Reduced Ejection Fraction (HFrEF) who have improved on the echocardiogram to an ejection fraction above 50%, patients with a previous ejection fraction between 40-49% who have progressed to ejection fraction above 50%. For these groups there is no need to perform the score for heart failure with preserved ejetion fraction score (since the diagnosis of HF was already known). Patients with signs/symptoms of HFpEF, who present structural morphological changes such as left atrium enlargement or left ventricular hypertrophy (LVH).
* After recently undergoing the score for heart failure with preserved ejetion fraction score (H2FPEF), patients who present scores that place them at least at an intermediate probability of HFpEF would be eligible for entry into the study.
* Signing the consent form

Exclusion Criteria:

* Patient with type I DM
* Estimated glomerular filtration rate (eGFR), using the Chronic Kidney Disease Epidemiology (CKD EPI) equation, with a cutoff of <20 mL/mm/1.73m2
* Patient currently using SGLT2 antagonists
* Patient with a history of allergic reaction or significant sensitivity to empagliflozin
* Female patient who is pregnant or considering becoming pregnant during the study or for 3 months after the last dose of study medication
* Patients that are breastfeeding
* Patients considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Patients with a previous diagnosis of HFpEF who presents a low probability of diagnosis after being re-stratified by the previously mentioned score
* Patients unable to walk or understand/comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Quality of life - application of Kansas City Cardiomyopathy Questionnaire | At inclusion and 60 days after receiving the medication.
  Applying the Kansas City Cardiomyopathy Questionnaire (KCCQ TSS) at inclusion and 60 days post-intervention in the two groups.
Quality of Life - Difference in the 6-minute walk test | At inclusion and 60 days after receiving the medication.
  Evaluate the difference in the 6-minute walk test before and after receiving the medication
Ejection fraction | Before receiving the drug and 60 days after.
  Using the echocardiogram upon entering the study, with assessment of ventricular and atrial strain modalities, repeating the same at the end of the treatment period to try to detect possible differences between pre and post treatment with the proposed Sodium-Glucose Transporter 2 Inhibitors (ISGLT2).

CONTACTS AND LOCATIONS:
Overall Officials: Conrado R Hoffmann Filho, Doctor, Principal Investigator — Multidisciplinary Center for Specialized Education and Research Ltd.
Locations (1):
- Multidisciplinary Center for Specialized Education and Research Ltd., Joinville, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No
Due to current Brazilian data protection law all individual participant data must be kept in secrecy.